CLINICAL TRIAL: NCT07218757
Title: A Pragmatic Trial of Emotional Awareness and Expression Therapy for Veterans With Chronic Pain: Phase 1
Brief Title: Phase 1 Pilot of a Pragmatic Trial of EAET for Veterans With Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); University of Texas Health Science Center at San Antonio (South Texas) ADRC (Unknown); University of Colorado, Denver (Other); University of Utah (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency); Yale University (Other); Greater Los Angeles Veterans Research and Education Foundation (Unknown)
Responsible Party: Principal Investigator, Brandon C. Yarns, MD, MS, BME, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1UG3AT013497-01 (NIH); 1UG3AT013497-01 (NIH)
Record Dates: First submitted 2025-10-16; First posted 2025-10-20 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Musculoskeletal Pain
Keywords: Chronic Pain; Psychotherapy; Musculoskeletal Disease; Mental Health
MeSH Terms: conditions — Musculoskeletal Pain; Chronic Pain; Musculoskeletal Diseases; Psychological Well-Being | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 either to emotional awareness and expression therapy (EAET) or cognitive behavioral therapy for chronic pain (CBT-CP). The randomization sequence will be generated at the start of the study by the study statistician using a computer randomizer to create seven sets of condition assignments (i.e., stratified by site) in blocks of 12 participants, resulting in 2 experimental groups of 6 participants after each block has been fully allocated. We consider 6 participants optimal because it is large enough to maintain group status even if someone drops out but small enough to provide individualized attention, facilitate scheduling a common group time, and keep the size of the pool to be randomized manageable.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Emotional awareness and expression therapy (EAET) (Experimental): Seeks to reduce physical (e.g., pain) and emotional (e.g., depression, anxiety) symptoms by helping individuals become aware of their emotions, express them, and resolve emotional conflicts. It will use techniques such as writing about stress, role playing how to handle difficult relationships, recognizing and expressing anger and other feelings, and being more open with others.
  Interventions: Behavioral: Emotional Awareness and Expression Therapy (EAET)
- Cognitive behavioral therapy for chronic pain (CBT-CP) (Active Comparator): Seeks to help individuals function better and improve symptoms by teaching various cognitive and behavioral skills to manage symptoms. It will use techniques such as relaxation training, engaging in pleasant activities, pacing yourself, and changing unhelpful ways of thinking.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Chronic Pain (CBT-CP)

INTERVENTIONS:
Behavioral: Emotional Awareness and Expression Therapy (EAET) — Talk therapy that helps people understand and express their feelings, especially emotions linked to past stress or trauma. The goal is to help reduce long-term pain by dealing with hidden emotional struggles that may be affecting the body.
  Arms: Emotional awareness and expression therapy (EAET)
Behavioral: Cognitive Behavioral Therapy for Chronic Pain (CBT-CP) — Talk therapy that helps people learn how their thoughts, feelings, and behaviors affect their pain. It teaches skills to manage pain, reduce stress, and improve daily life.
  Arms: Cognitive behavioral therapy for chronic pain (CBT-CP)

SUMMARY:
About one in three Veterans lives with long-term (chronic) pain, and many of them also struggle with past trauma and mental health issues like depression, anxiety, or PTSD. Emotional Awareness and Expression Therapy (EAET) is a type of talk therapy that helps people understand and express their emotions, especially those linked to past trauma. This therapy has been shown to help reduce pain and improve mental health.

So far, multiple studies have tested EAET in both Veterans and civilians, and the results have been promising. EAET has helped people feel less pain, move better, and experience fewer mental health symptoms. Because of these strong results, the U.S. Department of Health & Human Services named EAET a Best Practice for managing pain in 2019.

Two earlier studies at a VA hospital in Los Angeles found that EAET worked even better than another well-known therapy called cognitive behavioral therapy for chronic pain (CBT-CP) for older Veterans. However, those studies were done in tightly controlled settings. Now, researchers want to see if EAET works just as well when it's used in everyday healthcare settings, by different types of doctors and therapists.

This new project will happen in two parts, but we will only focus on the first part in this entry: In the first part (a 1-year phase), doctors and therapists at up to 7 VA hospitals across the country will be trained to use EAET. They will then try it out with Veterans to see how well it works and how easy it is to use in real clinics. Veterans, doctors, and other staff will be asked for feedback to learn what helps or gets in the way of using EAET.

DETAILED DESCRIPTION:
Chronic pain is present in nearly one-third of Veterans and is frequently accompanied by comorbid trauma and mental health symptoms. Emotional awareness and expression therapy (EAET) is an evidence-based psychological treatment for chronic pain that was developed to directly target comorbid trauma and mental health symptoms with the goal of reducing or eliminating chronic pain. Multiple controlled and uncontrolled efficacy trials of EAET in Veterans and civilians have shown EAET can produce robust effects on improving outcomes that include pain severity, pain interference, depression, anxiety, and post-traumatic stress disorder (PTSD) symptoms. Consequently, EAET was recommended as a Pain Management Best Practice by the U.S. Department of Health & Human Services in 2019. Moreover, in two single-site efficacy trials conducted at VA Greater Los Angeles Healthcare System, EAET was found to be superior on several outcomes to gold- standard cognitive behavioral therapy for chronic pain (CBT-CP) among older Veterans with chronic pain. Yet these more tightly controlled trials may not reflect the true effectiveness of EAET when implemented by diverse clinicians. The overall goal of the proposed project is to conduct a rigorous and comprehensive evaluation of EAET delivered in usual care settings. The project will proceed in two phases, but this entry will focus on the first phase: During a 1-year UG3 phase, clinicians at up to 7 geographically diverse VA healthcare systems will be trained in EAET via an EAET learning collaborative, and a pilot randomized clinical trial of EAET and CBT-CP will be performed at each site to confirm feasibility. In addition, a formative evaluation will be conducted to engage clinicians, administrators, and Veterans and to identify barriers and facilitators to implementation.

ELIGIBILITY:
Inclusion Criteria:

* Veteran at one of 7 VA healthcare systems;
* Age 18 years or older;
* At least 3 months of musculoskeletal pain, defined using International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) diagnostic codes, which include the following M-code diagnoses: back pain, fibromyalgia, limb pain, neck pain; R-code diagnoses: pelvic and perineal pain, jaw pain; and G-code diagnoses: tension headaches; and
* Pain of at least moderate severity, defined as ≥4 "on average" on the 0-10 Numeric Pain Rating Scale

Exclusion Criteria:

* Poorly controlled major psychiatric illness (e.g., schizophrenia, bipolar I disorder with acute psychotic symptoms, severe manic or depressive episode listed as active in CPRS);
* Active suicide or violence risk (e.g., currently suicidal or homicidal ideation, intent, or plans);
* Active severe drug/alcohol use disorder (e.g., drinking more than intended, tried to stop but couldn't, spent significant time drinking or being sick from aftereffects, wanted drink so badly you couldn't think of anything else, interference with home or work life, continued to drink despite problems, given up on activities, dangerous situations, withdrawal and/or tolerance); and
* Current participation in CBT-CP or EAET, or participation in either intervention in the last 6 months, via clinical care or another research study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2026-01-02 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Change in "pain severity" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  Brief Pain Inventory (BPI) Pain Severity. Average of four self report items: current pain, worst pain over the last 7 days, least pain over the last 7 days, and average pain over the last 7 days. Each item is scored 0-10 (0 = no pain; 10 = pain as bad as can be).

SECONDARY OUTCOMES:
Change in "pain Interference" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  BPI Pain Interference. Average of seven self-report items: general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Each item is scored 0-10 (0 = does not interfere; 10 = completely interferes).
Change in "total pain impact" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  Pain, Enjoyment of Life and General Activity scale. Average of three self-report items: average pain intensity, interference with enjoyment of life, and interference with general activity over the past week. Each item is scored 0-10 (0 = no pain or no interference; 10 = pain as bad as you can imagine or completely interferes).
Change in "physical functioning" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  PROMIS Physical Functioning Short Form 6b. Total of six self-report items assessing ability to perform daily physical activities such as carrying groceries, climbing stairs, walking, and self-care. Each item is scored on a 5-point scale (1 = unable to do; 5 = without any difficulty), with higher scores indicating better physical functioning.
Change in "sleep" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  PROMIS Sleep Disturbance 6a. Total of six self-report items assessing perceptions of sleep quality, difficulty falling asleep, and sleep satisfaction over the past 7 days. Each item is scored on a 5-point scale (e.g., 1 = not at all; 5 = very much), with higher scores indicating greater sleep disturbance.
Change in "fatigue" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  PROMIS Fatigue 7a. Total of seven self-report items assessing the frequency and impact of fatigue over the past 7 days, including tiredness, energy level, and how fatigue interferes with daily activities. Each item is scored on a 5-point scale (e.g., 1 = not at all; 5 = very much), with higher scores indicating greater fatigue.
Change in "pain catastrophizing" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  Pain Catastrophizing Scale-Short Form-6 Item. Total of six self-report items assessing catastrophic thinking related to pain, including rumination, magnification, and helplessness. Each item is scored 0-4 (0 = not at all; 4 = all the time), with higher scores indicating greater pain catastrophizing.
Change in "depression symptoms" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  Patient Health Questionnaire-8 Item. Total of eight self-report items assessing symptoms of depression over the past 2 weeks, including mood, interest, sleep, energy, appetite, self-worth, concentration, and psychomotor changes. Each item is scored 0-3 (0 = not at all; 3 = nearly every day), yielding a total score between 0 and 24, with higher scores indicating more severe depressive symptoms.
Change in "anxiety symptoms" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  Generalized Anxiety Disorder Scale-7 Item. Total of seven self-report items assessing symptoms of generalized anxiety over the past 2 weeks, including nervousness, uncontrollable worry, excessive worry, trouble relaxing, restlessness, irritability, and fear of something awful happening. Each item is scored 0-3 (0 = not at all; 3 = nearly every day), yielding a total score between 0 and 21, with higher scores indicating more severe anxiety symptoms.
Change in "PTSD symptoms" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  PTSD Checklist for DSM-5 (PCL-5). Total of 20 self-report items assessing PTSD symptoms over the past month, including intrusion, avoidance, negative alterations in cognition and mood, and alterations in arousal and reactivity. Each item is scored 0-4 (0 = not at all; 4 = extremely), yielding a total score between 0 and 80, with higher scores indicating greater PTSD symptom severity.
Change in "substance use screener" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  Tobacco, Alcohol, Prescription Medication, and Other Substance use first stage screener (TAPS-1). Single self-report item assessing frequency of use for tobacco, alcohol, prescription medications, and other substances over the past 12 months or since the last assessment point. Each item is scored on a scale from 0 to 5 (0 = never; 5 = daily or almost daily), with higher scores indicating greater substance use frequency.
Change in "World Health Organization Quality of life" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  World Health Organization-Quality of Life (WHOQOL-2). Two self-report items assessing overall quality of life and general health. Each item is scored on a 5-point scale (e.g., 1 = very poor/very dissatisfied; 5 = very good/very satisfied), with higher scores indicating better quality of life.
"Patient Global Impression of Change" at 10 weeks, 6 months, and 12 months post baseline | 10 weeks, 6 months, and 12 months post baseline
  Patient Global Impression of Change (PGIC). A single self report item assessing the Patient Global Impression of Change as a result of treatment. Items range from 1-7 (1 = No change (or condition has gotten worse); 7 = A great deal better and a considerable improvement that has made all the difference).

OTHER OUTCOMES:
Change in "pain attributions" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  Chronic Pain Attributions Scale v2 Short Form. Six self-report items assessing beliefs about the causes and consequences of chronic pain, including factors such as controllability and permanence. Three items are open ended and ask for write-in of the three main causes of their pain. The other three items are individually scored on a Likert scale (e.g., 1 = strongly disagree; 5 = strongly agree), with higher scores reflecting stronger endorsement of specific pain attributions.
Change in "emotional processing" from baseline to 10 weeks, 6 months, and 12 months post baseline | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  Emotional Processing Scale-15. Total of 15 self-report items assessing difficulties in processing emotions across multiple domains, including suppression, avoidance, and unregulated emotional responses. Each item is scored on a 0-4 scale (0 = strongly disagree; 4 = strongly agree), with higher scores indicating greater problems with emotional processing.
Change in "kinesiophobia" from baseline to 10 weeks, 6 months, and 12 months post baseline. | Baseline, along with 10 weeks, 6 months, and 12 months post baseline
  Tampa Scale for Kinesiophobia-11. Total of 11 self-report items assessing fear of movement or re-injury related to physical activity. Each item is scored on a 4-point scale (1 = strongly disagree; 4 = strongly agree), with higher scores indicating greater kinesiophobia (fear of movement).

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided